CLINICAL TRIAL: NCT07405710
Title: Choice of Diction's Effect: Electronic Measures of Resuscitation Status Inpatient
Brief Title: Use of the Electronic Medical Record to Screen Code Status Preference Using Death Language
Acronym: CODE-EMRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Karthik Joshua Kota, MD MPH, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2025000307
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Code Status Discussions With Medical In-patients
Keywords: Code status; CPR; EMR; Death language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental/Death language (Experimental): Participants will be asked:
  The purpose of this trial is to understand how the words we use to describe CPR affect patient decisions. Cardiopulmonary resuscitation (CPR) is performed when the heart stops beating. It consists of electric shocks to the heart, pumping the chest to circulate blood, and using a breathing machine to help with breathing. The success rate of CPR is about 1 in 7, and even when the heart restarts, the brain and other organs can be damaged. If your heart were to stop beating and you were to die without resuscitation, would you prefer that we attempt cardiopulmonary resuscitation (CPR), or would you prefer that we do not resuscitate (DNR)?
  Interventions: Behavioral: Death language
- Standard/non-death language (No Intervention): Participants will be asked:
  The purpose of this trial is to understand how the words we use to describe CPR affect patient decisions. Cardiopulmonary resuscitation (CPR) is performed when the heart stops beating. It consists of electric shocks to the heart, pumping the chest to circulate blood, and using a breathing machine to help with breathing. The success rate of CPR is about 1 in 7, and even when the heart restarts, the brain and other organs can be damaged. If your heart were to stop beating, would you prefer that we attempt cardiopulmonary resuscitation (CPR), or would you prefer that we do not resuscitate (DNR)?

INTERVENTIONS:
Behavioral: Death language — We will explicitly mention death when letting the participant know about CPR
  Arms: Experimental/Death language

SUMMARY:
In order to systematically improve code status communication and documentation while clarifying how providers understand code status decisions, we propose the Choice of Diction's Effect Electronic Measures of Resuscitation Study Inpatient (CODE-EMRS.I) with 3 aims: Aim 1 - Determine rate of patient utilization of code status invitation (research) via the Portal (Hypothesis 1: Participants with an existing Portal are more likely to participate in research than new signups); Aim 2 - Evaluate different phrasings in code status prompts with and without death language (Hypothesis 2: Participants are more likely to pick no code with death language than without); Aim 3 - Determine how objective data drives physician agreement on code status decision (Hypothesis 3: Physicians are more likely to disagree with full code decisions for poor GO-FAR, but not CCI). Participants will fill out all study questionnaires electronically, but have options within these to ask to speak to a study physician/their own physician for clarification. After completing the surveys, the research associate will deliver the patient's code status decision to the attending of record and ask their views on it. Once a week, participants who have expressed interest in the study (by clicking the "I am interested" button) but have not completed the study will receive a reminder to complete the study as well as an offer to withdraw from the study in that same communication.

ELIGIBILITY:
Inclusion Criteria:

* Age >65, English-fluency in reading and speaking, and the capacity to consent

Exclusion Criteria:

* Requiring ICU-level care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Code status decision | At enrollment
Physician of record decision for and agreement with code status | Within 24 hours of patient decision

CONTACTS AND LOCATIONS:
Overall Officials: Karthik J Kota, MD MPH, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Robert Wood Johnson University Hospital - New Brunswick, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will be made available upon request to the Department of Medicine and approval of the data elements by appropriate regulatory elements in the Department